CLINICAL TRIAL: NCT00608868
Title: A Phase IV, Multicenter, Non-randomized, Open-labeled Study to Evaluate the Efficacy of Gefitinib (IRESSA®) as a Second-line Therapy in NSCLC Patients
Brief Title: SELINE: Second-Line Iressa Phase IV Study in NSCLC Patients
Acronym: SELINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7913L00067
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-08

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Carcinoma; Non Small Cell Lung; EGFR mutation; Gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Gefitinib tablet 250mg once daily orally

SUMMARY:
The purpose of this study is to evaluate ORR (Objective Response Rate) of gefitinib as a second-line therapy for NSCLC patients based on RECIST (Response Evaluation Criteria in Solid Tumors Group) and check up ORR difference by EGFR mutation, gender, smoking history, and type of tumor.

ELIGIBILITY:
Inclusion Criteria:

* Pathological Diagnosis of local advanced/metastatic Non Small Cell Lung Carcinoma
* Previously failed the first-line chemotherapy
* Patient who can provide sample for EGFR mutation test

Exclusion Criteria:

* Central Nervous System metastasis or spinal cord compression that has not yet been definitively treated with surgery and/or radiation
* Any evidence of clinically active interstitial lung disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Daegu, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2007 to July 2008, 156 subjects were enrolled from 11 centers in Korea. First subject in date: 17 January 2007. Last subject last visit(Data cut off) date: 2 January 2009.
Pre-assignment Details: The subjects were able to provide sample of EGFR mutation test and the subjects who had positive EGFR results or satisfy more than two condition of adenocarcinoma, female or non smoker were eligible.
Groups:
- Gefitinib: gefitinib tablet 250 mg orally
Period: Overall Study
Arm/Group | Gefitinib
Started | 156
Enrolled | 156
Safety Population | 154 (2 patients who received no study treatment were excluded)
Treatment Completed | 141
Intention to Treat (ITT) Population | 138 (8 patients who had no target lesion and 8 who had no tumor assessment after baseline were excluded)
Per Protocol (PP) Population | 121
Completed | 141
Not Completed | 15
Not completed — Withdrawal by Subject | 7
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gefitinib
Number analyzed (Participants) | 138
Age, Customized [Number; unit: participants]
  < 65 years | 72
  >= 65 years | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 18
EGFR mutation status [Number; unit: Participants] — Epidermal growth factor receptor (EGFR) mutation analysis, PCR test on exon 18, 19 and 21 of EGFR gene was used.
  Participants
    Positive | 59
    Negative | 50
    Unknown | 29
Smoking history [Number; unit: Participants]
  Never-smoker | 117
  Ex-smoker | 17
  Regular smoker | 4
Tumour history [Number; unit: Participants]
  Adenocarcinoma | 121
  Squamous carcinoma | 13
  Other | 4
World Health Organisation (WHO) Performance Status [Number; unit: Participants] — WHO has 5 grades (0-4), 0 -Fully active, 1-Restricted in strenuous activity, 2- Ambulatory and capable of all self-care, 3-Capable of only limited self-care and 4- Completely disabled.
  Participants
    0 | 50
    1 | 73
    2 | 15
Disease Stage [Number; unit: Participants] — The tumor node metastasis (TNM) staging system (NSCLC) was used to determine the disease stage. Stage is usually expressed as a number on a scale of 0 through IV - with stage 0 describing non-invasive cancers that remain within their original location and stage IV describing invasive cancers that have spread outside to other parts of the body. Number of patients with different disease stage is reported.
  Participants
    I | 1
    III A | 4
    III B | 20
    IV | 113

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate(ORR)
Description: Primary efficacy endpoint is a change in the proportion of subjects showing overall objective response rate(ORR) from baseline to final tumor assessment point after treatment. As per RECIST, the percentage of subjects indicating PR (partial response) or CR (complete response) will be calculated.
  According RECIST criteria, CR(complete response) - the disappearance of all target lesions and 'PR(partial response) - at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: Every 8 weeks until progression disease or death or Data Cut off date (2 January 2009)
Measure: Number; unit: Percent of participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 138
Percent of participants | 31.2

2. Secondary Outcome: Period of Progression-Free Survival
Description: The median months without event of progression disease according to RECIST criteria is analysed.
Time Frame: Every 8 weeks until progression disease or death or Data Cut off date (2 January 2009)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gefitinib
Number analyzed (Participants) | 138
months | 5.7 [3.9 to 8.4]

3. Secondary Outcome: Quality of Life and Symptom Improvement Based on Functional Assessment of Cancer Therapy-Lung (FACT-L)
Description: Patients recorded the presence and severity of 7 symptoms by using the lung cancer subscale(LCS) at FACT-L; shortness of breath, weight loss, clarity of thinking, cough, appetite, chest tightness, and difficulty breathing. Severity was assessed by using 0~4 scale (0=not at all to 4=very much). A possible score was 0~28.
  The improvement rate defined as change of ≥6 points in overall FACT-L from baseline and the rate of patients who reported the change of points ≥2 in LCS of FACT-L.
  The percentage of patients who showed improvement is reported.
Time Frame: Every 8 weeks until progression disease or death or Data Cut off date (2 January 2009)
Measure: Number; unit: percentage of participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 94
percentage of participants | 41

4. Secondary Outcome: Overall Survival
Time Frame: Every 8 weeks until progression disease or death or Data Cut off date (2 January 2009) and every 12 weeks after progression until death or death.
Reporting Status: Not Posted
Measure: Number; unit: month

5. Secondary Outcome: Adverse Event
Description: An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Time Frame: Every 8 weeks until progression disease or death or Data Cut off date (2 January 2009)
Measure: Number; unit: participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 154
participants | 141

ADVERSE EVENTS:
Description: An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Arm/Group | Gefitinib
Serious Adverse Events (participants affected / at risk) | 25/154
Other Adverse Events (participants affected / at risk) | 141/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (N=154)
Cardiac tamponade (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Asthenia (Gastrointestinal disorders) | 2
Death (Gastrointestinal disorders) | 3
Multi-organ failure (Gastrointestinal disorders) | 1
Sudden death (Gastrointestinal disorders) | 1
Empyema (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (N=154)
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 40
Vomiting (Gastrointestinal disorders) | 8
Asthenia (Gastrointestinal disorders) | 12
Chest pain (Gastrointestinal disorders) | 10
Upper respiratory tract infection (Infections and infestations) | 13
Anorexia (Metabolism and nutrition disorders) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 27
Rash (Skin and subcutaneous tissue disorders) | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less